CLINICAL TRIAL: NCT06205095
Title: A Multi-cEnter, Pilot, Crossover Trial of Prophylactic Wilate CoMpared to PlacebO for Heavy Menstrual Bleeding in Patients with Von WillEbRand Disease
Brief Title: A Pilot Crossover Trial of Prophylactic Wilate Compared to Placebo for Heavy Menstrual Bleeding in Patients with VWD
Acronym: EMPOWER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2.5
Record Dates: First submitted 2023-12-18; First posted 2024-01-12 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Von Willebrand Diseases
MeSH Terms: conditions — von Willebrand Diseases | interventions — Factor VIII; von Willebrand Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pdVWF:FVIII concentrate (Wilate®) Treatment and Standard Care (Experimental): Wilate® at a dose of 30-60 IU VWF:RCo/kg for the two anticipated heaviest days of bleeding every 24-48 hours within the first 4 days of menstruation will be provided. Additional two optional doses 24-48 hours from the last can be provided. A minimum of 2 doses must be provided.
  Interventions: Drug: Lyophilized concentrate of human coagulation von Willebrand Factor and factor VIII
- Placebo and Standard Care (Placebo Comparator): Patients randomized to the placebo arm will receive intravenous placebo (normal saline) at the same approximate volume and frequency as the study drug.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lyophilized concentrate of human coagulation von Willebrand Factor and factor VIII — Wilate® is a plasma-derived, highly purified concentrate administered through intravenous injection. Wilate® contains an average VWF ristocetin cofactor activity to FVIII activity at ratio of 1:1.
  Other Names: Wilate
  Arms: pdVWF:FVIII concentrate (Wilate®) Treatment and Standard Care
Other: Placebo — Patients randomized to the placebo arm will receive intravenous normal saline at the same approximate volume and frequency of Wilate ®.
  Arms: Placebo and Standard Care

SUMMARY:
The EMPOWER trial is a pilot multi-center, placebo-controlled (normal saline), double-blind (patient and outcome assessor), crossover, 2-year randomized trial in female outpatients with von Willebrand disease (VWD) and heavy menstrual bleeding to determine trial feasibility and viability, and to explore assay sensitivity of the proposed efficacy clinical outcomes for a definitive randomized controlled trial

DETAILED DESCRIPTION:
The EMPOWER trial is a pilot multi-center, placebo-controlled (normal saline), double-blind (patient and outcome assessor), crossover, 2-year randomized trial in female outpatients with von Willebrand disease (VWD) and heavy menstrual bleeding to determine trial feasibility and viability, and explore assay sensitivity of the proposed efficacy clinical outcomes for a definitive randomized controlled trial.

For the first treatment period, patients will be randomized to receive either plasma derived von Willebrand factor:Factor VIII (pdVWF:FVIII) concentrate (plus standard of care) or placebo (plus standard of care) for VWD-associated heavy menstrual bleeding for 4 cycles, crossing over to the comparator treatment during the second treatment period. The first treatment period will be followed by a 1 cycle washout period when no study-based treatment will be delivered.

The main purpose of the pilot will be to evaluate viability and feasibility of the trial design, as well as to explore assay sensitivity to inform determination of the primary efficacy outcome for the definitive randomized trial which will evaluate the effect of prophylaxis with pdVWF:FVIII concentrate compared with placebo on HMB in women with VWD. A secondary objective is to conduct a preliminary assessment of the effect on clinical outcomes of 2-3 doses of prophylaxis with pdVWF:FVIII concentrate when provided on the first 4 days of menstruation compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patient capable of providing informed consent;
2. Female patients with HMB over the age of 18 years, for whom prophylactic treatment with Wilate® is deemed clinically appropriate according to the medical discretion (based on their expert opinion given consideration of the patient's bleeding history and responsiveness to treatment) of the treating hemostasis-focused physician practicing at a Hemophilia Treatment Center;
3. Modified PBAC score > 100 at screening;
4. Patients with a diagnosis of inherited von Willebrand disease (any type);
5. Stable treatment for HMB and iron deficiency anemia for 3 cycles before entering the study and anticipated to remain unchanged for the duration of the study;
6. Patients willing to have an infusion administered by a nurse over the course of the study period;
7. Patients who agree to use only the feminine hygiene products supplied by the sponsor.

Exclusion Criteria:

1. Diagnosed with any other known bleeding disorder;
2. Pregnancy or plans to become pregnant within the duration of the study;
3. Breastfeeding or plans to breastfeed within the duration of the study;
4. Known hypersensitivity reactions to human plasma-derived products or any ingredient in the formulation;
5. Known antibodies to VWF or FVIII;
6. Severe liver disease;
7. Anticipated initiation of the following: oral, transdermal, injectable, and vaginal ring hormonal contraceptives; GnRH analogues; or a hormonal intrauterine device (IUD) within the study period;
8. Anticipated elective procedure that is expected to require intensive treatment with VWF or FVIII for >10 days during the study period;
9. Patients with >2 risk factors for VTE (risk factors are determined at discretion of treating physician) or recent history of thrombosis (i.e. within the last year).
10. Patient concurrently receiving desmopressin (desmopressin cannot be taken concurrently with Wilate®, except for in the context of escalation treatment for excessive bleeding).
11. Anticipated initiation of any new therapies for the treatment of heavy menstrual bleeding 3 weeks prior to enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Blinding Index (BI) score at the end of cycle 4 of treatment period 1 and 2 | 2 years
  Blinding Index (BI) score at the end of cycle 4 of treatment period 1 and 2
Proportion of participant drop-out at the end of treatment period 1 and 2 | 2 years
  Proportion of participant drop-out at the end of treatment period 1 and 2
Proportion of participants with completed for the candidate primary clinical efficacy outcomes at the end of treatment period 1 and 2 | 2 years
  Proportion of patients with completed for the candidate primary clinical efficacy outcomes at the end of treatment period 1 and 2
Number of participants enrolled in 2 years (i.e. ability to enroll at least 10 participants in 2 years) | 2 years
  Ability to enroll at least 10 participants in 2 years
Proportion of participants with carryover effect for the candidate primary clinical efficacy outcomes from period 1 to period 2 | 2 years
  Proportion of participants with carryover effect for the candidate primary clinical efficacy outcomes from period 1 to period 2

SECONDARY OUTCOMES:
Mean of the 3 highest daily Modified PBAC (mPBAC) scores within each individual participant cycle averaged across 4 individual participant cycles at the end of each treatment period | At the end of 8 menstrual cycles (approximately 10 days)
  Mean of the 3 highest daily Modified PBAC (mPBAC) scores within each individual participant cycle averaged across 4 individual participant cycles at the end of each treatment period
The proportion of patients who use of rescue therapy at the end of each treatment period | At the end of 8 menstrual cycles (approximately 10 days)
  The proportion of patients who use of rescue therapy (i.e. more than two days of oral tranexamic acid use, additional treatment with Wilate®, additional hormonal therapy for HMB, urgent/emergent gynecological surgery for HMB, treatment with intravenous iron, red blood cell transfusion, or hospital admission for HMB) at the end of each treatment period
Mean of the mPBAC score within each individual participant cycle averaged across 4 individual participant cycles | At the end of 8 menstrual cycles (approximately 10 days)
  Mean of the mPBAC score within each individual participant cycle averaged across 4 individual participant cycles
Median of the mPBAC score within each individual participant cycle used to derive the median across 4 individual participant cycles | At the end of 8 menstrual cycles (approximately 10 days)
  Median of the mPBAC score within each individual participant cycle used to derive the median across 4 individual participant cycles
Number of days of oral tranexamic acid use | At the end of 8 menstrual cycles (approximately 10 days)
  Number of days of oral tranexamic acid use
Number of days of Wilate® treatment received | At the end of 8 menstrual cycles (approximately 10 days)
  Number of days of Wilate® treatment received
Duration of menstruation (measured in days) | At the end of 8 menstrual cycles (approximately 10 days)
  Duration of menstruation (measured in days)
Major bleed according to the International Society on Thrombosis and Haemostasis (ISTH) definition | At the end of 8 menstrual cycles (approximately 10 days)
  Major bleed according to the International Society on Thrombosis and Haemostasis (ISTH) definition
Clinically relevant non-major bleed | At the end of 8 menstrual cycles (approximately 10 days)
  Clinically relevant non-major bleed
Hemoglobin levels (g/L) | At the end of 8 menstrual cycles (approximately 10 days)
  Hemoglobin levels (g/L)
Ferritin levels (mcg/L) | At the end of 8 menstrual cycles (approximately 10 days)
  Ferritin levels (mcg/L)
Use of additional hormonal therapy for heavy menstrual bleeding | At the end of 8 menstrual cycles (approximately 10 days)
  Use of additional hormonal therapy for heavy menstrual bleeding
Requirement of urgent/emergent gynecological surgery for heavy menstrual bleeding | At the end of 8 menstrual cycles (approximately 10 days)
  Requirement of urgent/emergent gynecological surgery for heavy menstrual bleeding
Fatigue scores (as measured by the FACIT fatigue scale) | At the end of 8 menstrual cycles (approximately 10 days)
  Fatigue scores (as measured by the FACIT fatigue scale)
Short Form-12 Scores | At the end of 8 menstrual cycles (approximately 10 days)
  Short Form-12 Scores
Scores on the individual components of the Short Form-12 | At the end of 8 menstrual cycles (approximately 10 days)
  Scores on the individual components of the Short Form-12
Requirement of hemostatic care (tranexamic acid, Wilate®, platelet transfusion) | At the end of 8 menstrual cycles (approximately 10 days)
  Requirement of hemostatic care (tranexamic acid, Wilate®, platelet transfusion)
Requirement of anemia focused care (intravenous iron and/or red blood cell transfusion) | At the end of 8 menstrual cycles (approximately 10 days)
  Requirement of anemia focused care (intravenous iron and/or red blood cell transfusion)
Number of hypersensitivity infusion reactions | At the end of 8 menstrual cycles (approximately 10 days)
  Number of hypersensitivity infusion reactions
Number of thromboembolic events (defined as symptomatic or incidental, suspected or confirmed via diagnostic imaging and/or electrocardiogram where appropriate); | At the end of 8 menstrual cycles (approximately 10 days)
  Number of thromboembolic events (defined as symptomatic or incidental, suspected or confirmed via diagnostic imaging and/or electrocardiogram where appropriate);
Proportion of participants who development of VWF inhibitors | At the end of 8 menstrual cycles (approximately 10 days)
  Proportion of participants who development of VWF inhibitors
Number of adverse events | 8 cycles
  Number of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No